CLINICAL TRIAL: NCT05529017
Title: Performance Characteristics and Post-injury Deficits in Rink Field Hockey
Brief Title: Post Injury Performance Deficits in Rink Hockey
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Hugo Olmedillas Fernandez, Associate professor, University of Oviedo
Other Study IDs: UO2022-03
Record Dates: First submitted 2022-07-25; First posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Injuries; Sports Physical Therapy; Non Contact Injury; Performance
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non/injured players: rink hockey players participating in senior leagues

SUMMARY:
Rink Hockey is a sport played on a 40*20 metres rink characterized by combined periods of high intensity and short breaks, there´s a lack of epidemiological studies in this field. In line with the well-established model of sports injury prevention research proffered by van Mechelen, the first stage in this process is establishing the extent of the problem i.e. injury incidence, severity and burden.

DETAILED DESCRIPTION:
This study will assess performance metrics from rink hockey athletes and injury epidemiology. 4 tests (to be specified yet) will evaluate players fitness during preseason and when a player suffers a non-contact injury during the season, the player will be retested to assess variability and performance deficits.

injury characteristics and exposure time will be recorded too

ELIGIBILITY:
Inclusion Criteria:

* Compete in senior league
* be uninjured during preseason

Exclusion Criteria:

* not signing the participation consent
* no participation in the performance assessment during preseason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: rink hockey players (male and female) from spanish senior leagues only outfield players irrespective of category
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Maximal strength capacity | september 2022 to june 2023
  The RM maximal resistance for the squat exercise will be estimated by performing the squat exercise with different weights and measuring barbell movement speed. Measuring the barbell speed we can estimate the 1RM since it follows a linear relationship with the weight the athlete must lift. Therefore, the higher the weight, the slower the barbell will be moved. 1RM is considered the weight moved at .2m/s by the participant.The value will be expressed in kilograms
injury incidence | september 2022 to june 2023
  number of injuries observed during the season 2022-2023
Explosive strength test (Countermovement jump test) | september 2022 to june 2023
  capacity of the athlete to display lower body explosive strength. it is measured with a slow motion camera and the app MyJump. The result is expressed in cm.
  The athlete performs a vertical jump as fast as possible with their hands around their waist
Agility test (5-10-5 test) | september 2022 to june 2023
  agility test for the lower body. three cones separated by 5 metres each. the participant starts in the middle cone, runs to one edge (5 metres) and then brakes and runs to the other (10 metres) to brake again and come back to the middle cone. the result is expressed in seconds that the participant needs to complete the test. the test is performed in skates.
cardiovascular fitness test (30-15 test) | september 2022 to june 2023
  this test aims to assess cardiovascular capacity of the athlete. the athlete runs at a certain pace (marked by an audio) along a 28m track. every time there is a beep the athlete must have completed the corresponding distance. every 30 seconds the speed increases and therefore the athlete must run faster. the result is the last speed the participant was skating at. when the participant fails to reach the corresponding distance 3 times, gets eliminated

SECONDARY OUTCOMES:
region injured | september 2022 to june 2023
  which body region was injured (lower limb only) according to the International Olympic Committee consensus statement
tissue affected | september 2022 to june 2023
  Injuries can affect different tissues in the body. The International Olympic Committee differs between muscle, ligament, tendon, nerve or bone injuries (among others: skin or central nervous system). Tissue injured will be analyzed to assess wether a certain tissue is more predisposed to getting injured than others.
injury burden | september 2022 to june 2023
  lay-off days due to the injury
mechanism of injury | september 2022 to june 2023
  Injuries can be cathegorized between contact and non-contact, in this study only non-contact lower body injuries will be analyzed. This information will be collected to assess which gesture provoked the injury (sprint, side brake, etc) and evaluate which specific movement is more injurious in this sport

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Olmedillas, PhD, Principal Investigator — Universidad de Oviedo

IPD SHARING:
Plan to Share IPD: No